CLINICAL TRIAL: NCT01641341
Title: Irritable Bowel Syndrome Evaluation and Treatment in Primary Care
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: American Academy of Family Physicians (Other)
Collaborators: Genova Diagnostics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 10-108
Record Dates: First submitted 2011-05-09; First posted 2012-07-16 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome; Genova Diagnostics kit; Stool test; Rome III; Practice-based research; treatable parasite; Pancreatic insufficiency; Bowel dysbiosis; High levels of inflammation, C. difficile, or H. pylori
MeSH Terms: conditions — Irritable Bowel Syndrome; Exocrine Pancreatic Insufficiency | interventions — bifidus factor; Probiotics; Pancrelipase; nitazoxanide; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo capsule (Placebo Comparator): Placebo capsule (sugar pill with no active medication)
  Interventions: Drug: Placebo
- Active treatment (Active Comparator): Active treatment will consist of the following interventions:
  1. Bowel Dysbiosis - probiotics Bifidobacterium infantis,
  2. Maldigestion/Malabsorption - Pancrelipase
  3. Parasitic infection/presence - Nitazoxanide
  Interventions: Drug: Bifidobacterium infantis; Drug: Pancrelipase; Drug: Nitazoxanide

INTERVENTIONS:
Drug: Bifidobacterium infantis — once a day for seven to eight weeks
  Other Names: B. Bifidum; B. Breve; B. Infantis; Bifidobacterias; Bifidobacterium bifidum; Bifidum; Bifidus; Probiotic
  Arms: Active treatment
Drug: Pancrelipase — Pancrelipase (one capsule prior to meals or snacks)
  Other Names: Lipancreatin
  Arms: Active treatment
Drug: Nitazoxanide — Nitazoxanide (500mg twice a day for 7 days)
  Other Names: Alinia
  Arms: Active treatment
Drug: Placebo — Placebo capsule will not contain active treatment ingredients.
  Other Names: Sugar pill
  Arms: Placebo capsule

SUMMARY:
Overview of Methods: This is a double blind, randomized controlled trial with a non-balanced randomization and a cross-over to active treatment for placebo treated individuals who do not respond to the placebo treatment. Data collected will help determine the feasibility of the study design in primary care offices. Patient outcome data will provide a more precise estimate of power for a larger, classic randomized trial to determine if such a study can be reasonably undertaken within primary care practices.

Aims: The aims of this pilot study are to: 1) Evaluate how well Genova Diagnostics (GDx) IBS tests can be integrated into primary care, 2) examine the effects of the Genova Diagnostics (GDx) test on treatment, and 3) observe and track patients' health, quality of life and clinical outcomes related to IBS during the study period.

DETAILED DESCRIPTION:
This study will take place in 8 practices which are members of the AAFP NRN. Eligible practices must be able to identify at least 25 active patients (seen in last 24 months) with a diagnosis of IBS from billing or electronic health record data to be eligible to participate. Each practice will be asked to recruit 10 patients.

Adult patients identified by their physician as having IBS symptoms will be termed "potentially eligible patients" and will be invited into the study via personal invitation when presenting at the practice on a regularly-scheduled visit, by letters mailed to these patients on practice letterhead and signed by the physician, or through phone contact with a member of the practice.

If a patient agrees to participate in the study, s/he will be asked to read and sign an initial informed consent. Consent forms will be included with the letters mailed to patients, and additional copies of the consent will be kept at the practice. The initial informed consent will cover consent for stool testing, for collection of all study outcome data including new diagnoses uncovered by the stool testing and any follow up procedures that are conducted as a result of the stool test results. This initial consent will indicate that based on stool testing results the patient may be referred for more evaluation or open label treatment from their physician or may be recommended for one or more study directed treatment(s).

Once the stool tests have returned the patient will be contacted to review these results. At that time the patient will be asked to sign a secondary consent form if study directed therapy is recommended. This consent form or these consent forms (if more than one therapy is recommended) will be treatment specific and explain that the patient will be randomized to active or placebo treatment in a double blinded fashion, that the patient will be crossed over to either active treatment or placebo after 8 weeks and that all patients will be offered active treatment by the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 18 and 65 years of age
* meet Rome III criteria for IBS
* willing to complete surveys and daily symptom logs for three to four 14-day periods
* have positive symptoms for at least 3 days out of the 14 days of the baseline daily log records

Exclusion Criteria:

* have HIV or AIDs
* have gall stones with a gall bladder present

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2010-11; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
A reduction in IBS symptoms | 16 weeks
  20 to 40% of the control/placebo patients and approximately 70-75% of the treatment patients will experience a positive outcome as determined by both the daily log sheets and the modified Rome criteria administered at baseline, 8 and 16 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Evelyn Lewis & Clark, MD, MA, Principal Investigator — National Research Network; Wilson Pace, MD, Study Chair — National Research Network; Gerard Mullin, MD, Study Chair — Johns Hopkins School of Medicine
Locations (9):
- United States (9):
  - Torrance Clinical Research, Lomita, California
  - Overland Park Family Health Partners, Leawood, Kansas
  - American Academy of Family Physicians-National Research Network, Leawood, Kansas
  - Baton Rouge Family Practice, Baton Rouge, Louisiana
  - Family Medicine of SE Missouri, Sikeston, Missouri
  - Missouri Delta Physician Services, Sikeston, Missouri
  - Silver Sage Center for Family Medicine, Reno, Nevada
  - Raj Kachoria, Macedon, New York
  - Southwest Family Medicine Associates, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No